CLINICAL TRIAL: NCT03486717
Title: The Use of Virtual Reality Goggles on Patient Pain and Behavior in Pediatric Dentistry; a Pilot Study
Brief Title: The Use of Virtual Reality Goggles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Casey Goetz (Other)
Responsible Party: Sponsor-Investigator, Casey Goetz, Pediatric Dentistry Resident, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 201803829
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Control (Experimental): Study group that does not wear the virtual reality goggles. This group will serve as a control.
  Interventions: Device: Virtual reality goggles

INTERVENTIONS:
Device: Virtual reality goggles — Patients will act as their own control over two different dental appointments. One appointment will consist of wearing the virtual reality googles, the other appointment will be conducted without them. The goggles have a small screen inside of them along with headphones. This device will play an a movie or cartoon that will immerse the patient during treatment.

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of virtual-reality audio-visual distraction goggles on pain and behavior scores in a population of 8-12 year old dental patients receiving routine dental care in an outpatient clinical setting.

DETAILED DESCRIPTION:
All appointments will take place at the College of Dentistry Department of Pediatric Dentistry. The first day's appointment will consist of clinically-indicated cleaning, radiographs and treatment planning. Toward the end of the first appointment, the participant will wear the virtual reality goggles for 5 minutes, in order to become familiar with the device. During these 5 minutes, fluoride varnish will be applied. The application of the varnish would occur whether the participant is in the research or not.

At the second or third appointments, the goggles will be randomly used during the restorative treatment. Whether the participant uses the goggles at the second or third visit will be determined purely by chance, like flipping a coin. No nitrous oxide will be used, but local anesthesia will still be administered as standard. The participant will use a 1-10 scale at the end of each appointment to rate pain levels, and a research team member(the dental assistant) will assign a 1-4 scale value for behavior. The 1-10 scale will consist of the Wong-Baker Faces Pain Scale.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, no history of seizures or neurological disturbance, requires two quadrants of dentistry

Exclusion Criteria:

* History of dental anxiety

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Self-reported patient perception of pain | recorded immediately after each treatment session, during both the control visit and the experimental visit (patient acts as their own control)
  The patient will complete a self-reported pain scale known as the Wong-Baker Faces Pain Scale. This is a 1-10 pain scale that has correlating faces. A 1 indicates no pain, and correlates with a happy face. A 10 correlates with a crying face and indicates severe pain. A single number between 1-10 is selected to indicate the patient's pain.
Behavior of child | recorded immediately after each treatment session, during both the control visit and the experimental visit (patient acts as their own control)
  Behavior in terms of child cooperation will reported by an unbiased dental assistant using the Frankyl behavior scale. Behavior means the child listens to instructions and follows directions given by the clinician. This is a 1-4 scale, with 1 indicating extremely uncooperative behavior (crying, strong movement) and 4 indicating positive, cooperative behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Casey Goetz, DDS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No